CLINICAL TRIAL: NCT05386524
Title: Efficacy and Safety of Sintilimab and Bevacizumab Biosimilar Combined With Pegylated Liposomal Doxorubicin in Pretreated Metastatic Triple-negative Breast Cancer: a Single Arm Phase II Trial
Brief Title: Sintilimab and Bevacizumab Biosimilar Combined With PLD in mTNBC
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Fudan University (Other)
Responsible Party: Principal Investigator, Biyun Wang, MD, Professor, Fudan University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: YOUNGBC-18
Record Dates: First submitted 2022-05-18; First posted 2022-05-23 (Actual); Last update posted 2023-02-16 (Actual); Status verified 2023-02

CONDITIONS: Breast Cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — sintilimab; liposomal doxorubicin

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- SBP group (Experimental): sintilimab 200mg, ivgtt，d1， bevacizumab biosimilar 15mg/kg，ivgtt d1， pegylated liposomal doxorubicin 30mg/m2 d1，q3w
  Interventions: Drug: sintilimab; Drug: bevacizumab biosimilar; Drug: pegylated liposomal doxorubicin

INTERVENTIONS:
Drug: sintilimab — sintilimab 200mg, ivgtt，d1
Drug: bevacizumab biosimilar — bevacizumab biosimilar 15mg/kg，ivgtt d1
Drug: pegylated liposomal doxorubicin — pegylated liposomal doxorubicin 30mg/m2 d1，q3w

SUMMARY:
To evaluate the efficacy and safety of sintilimab and bevacizumab biosimilar combined with pegylated liposomal doxorubicin in pretreated metastatic triple-negative breast cancer

ELIGIBILITY:
Inclusion Criteria:

* Patients aged 18-70 years old.
* Metastatic breast cancer included unresectable locally advanced breast cancer, de novo stage IV breast cancer, and recurrent metastatic breast cancer.
* ER and PR negative, HER2 negative breast cancer.
* Received one or two lines of systemic treatment in metastatic setting
* Measurable disease based on RECIST 1.1.
* ECOG Performance Status 0-1
* Adequate hematological, renal and hepatic function according to all of the following laboratory values

Exclusion Criteria:

* Has received any prior therapy with an anti-PD-1, anti-PD-L1, or anti-PD-L2 agent
* Has received any prior therapy with bevacizumab.
* Has a diagnosis of immunodeficiency or is receiving chronic systemic steroid therapy (in dosing exceeding 10 mg daily of prednisone equivalent)
* Has a known additional malignancy that is progressing or has required active treatment within the past 5 years with the exception of basal cell carcinoma of the skin, squamous cell carcinoma of the skin, or carcinoma in situ (eg, cervical cancer in situ) that have undergone potentially curative therapy
* Has known active central nervous system (CNS) metastases and/or carcinomatous meningitis
* Has a known history of hypersensitivity (≥ Grade 3) to pembrolizumab and/or any of its excipient
* Has an active autoimmune disease that has required systemic treatment
* Has a history of (non-infectious) pneumonitis that required treatment with steroids; or current pneumonitis.
* Has a history or current evidence of any condition, therapy, or laboratory abnormality that might confound the results of the study, interfere with the participant's participation for the full duration of the study, or is not in the best interest of the participant to participate, in the opinion of the treating investigator.
* Has a known psychiatric or substance abuse disorder that would interfere with the participant's ability to cooperate with the requirements of the study
* Has been pregnant or breastfeeding or expecting to conceive or father children within the projected duration of the study, starting with the screening visit through 180 days after the last dose of trial treatment.
* Failure to comply with the study procedures, restrictions and requirements of the study

Ages: 18 Years to 70 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 41 (Estimated)
Dates: Start 2022-06-15 (Actual); Primary Completion 2025-03-15 (Estimated); Study Completion 2025-03-15 (Estimated)

PRIMARY OUTCOMES:
PFS | 6 weeks
  Progression free survival
OS | 6 weeks
  Overall Survival
Adverse Events | 6 weeks
  Number of participants with treatment-related adverse events as assessed by CTCAE v 5.0

CONTACTS AND LOCATIONS:
Overall Officials: Biyun Wang, Prof, Principal Investigator — Fudan University
Locations (1):
- Fudan University Shanghai Cancer Center, Shanghai, Shanghai Municipality, China